CLINICAL TRIAL: NCT04194827
Title: Adalimumab Drug Optimisation in Rheumatoid Arthritis Using Therapeutic Drug Monitoring (ADDORA): Multi-centre Open Label Randomised Controlled Trail
Brief Title: Adalimumab Drug Optimisation in Rheumatoid Arthritis Using Therapeutic Drug Monitoring
Acronym: ADDORA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Reade Rheumatology Research Institute (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADDORA
Record Dates: First submitted 2019-12-03; First posted 2019-12-11 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Adalimumab; Rheumatoid arthritis; Therapeutic Drug Monitoring; Drug level; Dose reduction
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: Rheumatoid arthritis patients treated with adalimumab will be randomly assigned to a dose reduction strategy using disease activity scores or to a dose reduction strategy using serum drug concentrations
Who Masked: Outcomes Assessor
Masking Description: During every study visit the joints of all patients will be examined for pain and swelling by a blinded nurse or physician. The number of painful and swollen joints will be used to calculate the DAS28 score, the primary outcome of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concentration guided dose reducion (Experimental): Dose reduction of adalimumab will be based on adalimumab through concentration after 16 weeks of treatment with adalimumab.
  Interventions: Diagnostic Test: Adalimumab serum trough concentration; Drug: Adalimumab
- Disease activity quided dose reduction (Active Comparator): Dose reduction of adalimumab will be based on disease activity after 28 weeks of treatment with adalimumab
  Interventions: Diagnostic Test: Disease activity; Drug: Adalimumab

INTERVENTIONS:
Diagnostic Test: Adalimumab serum trough concentration — Dose reduction based on adalimumab serum trough concentration
  Arms: Concentration guided dose reducion
Diagnostic Test: Disease activity — Dose reduction based on adalimumab diseas activity
  Arms: Disease activity quided dose reduction
Drug: Adalimumab — Adalimumab

SUMMARY:
Several prior studies have shown that dose reduction of Tumor Necrosis Factor (TNF)-inhibitors like adalimumab is possible in substantial number of rheumatic disease patients without an increase in disease activity. Biologic therapy is expensive, and is associated with patient burden as dose dependant risk for serious infections . A dose reduction will decrease the risk of side effects and result in substantial cost savings. Currently, most clinicians use Disease Activity Score in 28 joints (DAS28) and the Clinical Disease Activity Index (CDAI) to monitor dose tapering strategies. Although this approach is cost-effective, it might be improved by information on the extent of drug levels, as several studies have shown that adalimumab drug levels are associated with clinical outcome. Therefore, a study comparing dose reduction strategy using drug concentration with dose reduction strategy using disease activity is timely

DETAILED DESCRIPTION:
Since the introduction of biologics in rheumatology, as well as treat-to-target (measuring disease activity and adapting treatment accordingly) the prognosis of patients has improved substantially. Obviously, patient burden due to self-injection or infusion, the risk of adverse events and costs demand responsible use of these agents. Multiple studies have shown that a large proportion of patients with rheumatoid arthritis with stable low disease activity can taper their dose or stop without relapse of disease activity. This can be done by using disease activity guided tapering. Drawbacks, however, include increased risk for short lived flares, the effort of slowly and carefully tapering, and somewhat more risk of radiographic damage due to higher mean disease activity. As most biologics are characterized by wide variation in pharmacokinetics between patients, therapeutic drug monitoring (TDM), i.e. dose based on serum trough concentration, might be an attractive approach to lower the dose quickly while remaining clinical efficacy. Although some data suggest that the minimal effective concentration varies between patients, we demonstrated in an earlier study that serum adalimumab concentration of 5 mg/L is enough for initial response to adalimumab. In the first phase of treatment, drug concentration must be high enough to control immunogenicity. To control disease activity after 28 weeks, lower concentrations than 5 mg/L are probably sufficient. Since around 70% of the patients have an adalimumab concentration above 5 mg/l, we assume that dose reduction to achieve these lower targets (for example direct doubling of interval in patients with levels > 10 mg/L) will result in the lowest effective drug dose. Our study group illustrated in 2018 that dose reduction by extending the dosing interval with 50% is non inferior to continuation of standard dose in patients with adalimumab levels > 8mg/L. In other words, measuring drug concentrations can help clinicians to select overexposed patients to reduce the dose of adalimumab without adversely affecting clinical efficiency. We posit that therapeutic drug monitoring can attribute to a more efficient dose reduction strategy. Since steady state drug concentrations are achieved within 16 weeks of treatment, we expect that the dose can be reduced from this point. This is earlier in treatment compared to the strategy using disease activity alone, namely after 6 months of treatment. Conceptually, such a test can improve disease activity guided dose reduction in two ways: 1) flaring caused by empirical tapering (i.e. through trial and error) below the minimal effective concentration would be avoided, and 2) patients can be directly given their minimum effective dose instead of empirical tapering, thereby saving time and drugs. Our aim is to investigate whether the use of drug levels can attribute to a more efficient dose reduction strategy of adalimumab in patients with RA. In this study we will compare costs and clinical efficiency of two dose reduction strategies: a strategy using drug concentration versus a strategy using disease activity scores. We expect that direct medical costs will be lower in the 'drug concentration guided' strategy because: 1) overexposed patient can reduce the dose more timely and, 2) adalimumab dose can be further reduced after 6 months of treatment since we posit that adalimumab concentration of 2 mg/L is sufficient to control disease.

In this multi-centre, randomised, open-label trail we will evaluate whether dose reduction of adalimumab using drug concentration can reduce medical costs compared to a strategy using disease activity scores. Furthermore we will evaluate the clinical efficiency of these two strategies.

Patients with a good or moderate EULAR response to adalimumab will be randomised to adalimumab dose reduction strategy using drug concentration or disease activity scores. Patients in the 'drug concentration guided' group will reduce adalimumab dose by prolonging the dose-interval using TDM algorithm (a new developed algorithm is used to determine the interval prolongation for each patient). The dose reduction will start at week 16 if trough drug level is higher than 5mg/L, aiming a drug level of 5mg/L in week 16 until 28 and a drug level of 2mg/L from week 28 until week 52. In the initial 16 weeks patients are treated with adalimumab at registered dose of 40mg every other week.

Patients in the 'disease activity guided' group will reduce adalimumab dose at week 28 if DAS28-CRP is lower than 2.9. This dose reduction will be attained by extending the dosing interval to every 3 weeks in weeks 28 until 40 and to every 4 weeks from week 40 until week 52.

Patients who successfully prolonged the dose interval to 40 mg every 4 weeks in the 'disease activity guided' group and patients who successfully prolonged their dose-interval and achieve a serum concentration of 2.0 mg/L in the 'drug concentration guided' group will be approached to participate to the extension phase (week 52-80). After informed consent is obtained patients will discontinue adalimumab and they will be followed up to week 80.

Data regarding disease status, functioning, adalimumab serum concentrations, anti-drug antibodies and medical costs will be collected during this study.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis patient, according to ACR 1987 or ACR/EULAR 2010 criteria;
* Starting adalimumab as the first biological therapy
* Who has agreed to participate (written informed consent);
* Age 18 years or older.

Exclusion Criteria:

* Scheduled surgery during the follow-up of the study or other pre-planned reasons for treatment discontinuation;
* Life expectancy shorter than follow-up period of the study;
* Other disease that might flare if adalimumab is tapered like psoriasis, inflammatory bowel disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Medical costs | 52 weeks
  Direct medical costs associated with adalimumab dose reduction using drug concentration versus using disease activity scores

SECONDARY OUTCOMES:
Mean time weighted DAS28-CRP | at 16, 28, 52 and 80 weeks
  Difference in mean time weighted DAS28-CRP
Direct medical costs | at week 28 and week 80
  Direct medical costs (medication, visits, cost TDM testing) at the separate time points
Indirect medical costs | at 28, 52 and 80 weeks
  Costs due to RA-related work absenteeism and presentism for patients with paid jobs and days of inactivity for patients without a paid job. Indirect costs will be estimated by three-monthly questionnaires, monitoring these items in the previous month (based on the SF-HLQ).
Patients with DAS28-CRP<2.9 | at 52 and 80 weeks
  Percentage of patients with DAS28-CRP<2.9
Number of flares | at 52 and 80 weeks
Number of dose-interval shortenings | at 52 and 80 weeks
Drug levels | at 4,16, 28, 40, 52 and 80 weeks
  The difference in drug levels between the measured drug level and the predicted drug level with the (newly developed) algorithm at different timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Gertjan Wolbink, PhD, Principal Investigator — Reade Rheumatology Research Institute
Locations (1):
- Reade Rheumatology Research Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
To avoid duplication of research, the gathered data will be shared once all desirable data analysis have been performed and the results are published
Supporting Information: Study Protocol, SAP
Time Frame: Six months after the study is published the data will be shared
Access Criteria: Researchers with demonstrable interest in autoimmunity, biologicals, or TDM can contact the investigators of the trial if they are interested in gaining access to the data. Depending on their research objectives the data will be shared

REFERENCES:
- [Background] Chen DY, Chen YM, Hsieh TY, Hung WT, Hsieh CW, Chen HH, Tang KT, Lan JL. Drug trough levels predict therapeutic responses to dose reduction of adalimumab for rheumatoid arthritis patients during 24 weeks of follow-up. Rheumatology (Oxford). 2016 Jan;55(1):143-8. doi: 10.1093/rheumatology/kev298. Epub 2015 Aug 31. PMID 26324949
- [Background] Kievit W, van Herwaarden N, van den Hoogen FH, van Vollenhoven RF, Bijlsma JW, van den Bemt BJ, van der Maas A, den Broeder AA. Disease activity-guided dose optimisation of adalimumab and etanercept is a cost-effective strategy compared with non-tapering tight control rheumatoid arthritis care: analyses of the DRESS study. Ann Rheum Dis. 2016 Nov;75(11):1939-1944. doi: 10.1136/annrheumdis-2015-208317. Epub 2016 Jan 13. PMID 26764260
- [Background] l'Ami MJ, Krieckaert CL, Nurmohamed MT, van Vollenhoven RF, Rispens T, Boers M, Wolbink GJ. Successful reduction of overexposure in patients with rheumatoid arthritis with high serum adalimumab concentrations: an open-label, non-inferiority, randomised clinical trial. Ann Rheum Dis. 2018 Apr;77(4):484-487. doi: 10.1136/annrheumdis-2017-211781. Epub 2017 Sep 22. PMID 28939629
- [Background] Pouw MF, Krieckaert CL, Nurmohamed MT, van der Kleij D, Aarden L, Rispens T, Wolbink G. Key findings towards optimising adalimumab treatment: the concentration-effect curve. Ann Rheum Dis. 2015 Mar;74(3):513-8. doi: 10.1136/annrheumdis-2013-204172. Epub 2013 Dec 10. PMID 24326008